CLINICAL TRIAL: NCT05632081
Title: Study of Asthma Step-up in Real Life (SURFE)
Brief Title: A Study of Step-up in Bronchial Asthma as a New End Point in Asthma Control (SURFE)
Acronym: SURFE
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hesham Raafat, A. professor chest medicine department, pulmonology consultant, Ain Shams University
Other Study IDs: SFHD001
Record Dates: First submitted 2022-11-19; First posted 2022-11-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Asthma step-up; Asthma step-down; Asthma exacerbation; Mild asthma; Moderate asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CBC, total IgE in some patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the frequency needed for stepping-up treatment in patients with mild and moderate bronchial asthma. The main questions this study aims to answer are:

* What is the frequency and duration in which patients of asthma need to step up their treatment?
* Can the criteria described in this study be applied and validated to test need for step up of asthma treatment? Participants will follow the treatment they are already receiving according to established guidelines and will be asked for regular visits for examination and spirometry. They will record symptoms score, each time they use the prescribed rescu inhaler, and morning and evening peak expiratory flow.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent.
2. Age above 12 years.
3. Ability to use study inhalers correctly, use e-diary, and comply with study procedures and visits.
4. Confirmed diagnosis of mild or moderate asthma asthma (based on GINA defined asthma control on a maximum of maintenance low dose ICS/LABA combination).
5. Pre-bronchodilator ≥FEV1 60%.
6. Reversibility test ≥12% or 200 ml from baseline.
7. Non-smoker.
8. For female subjects, non-pregnant and administer efficient contraception if in childbearing period.

Exclusion Criteria:

1. Severe asthma exacerbation in last 3 months.
2. Use of any systemic corticosteroids in last 12 weeks.
3. Use of depot systemic steroids in last 12 weeks.
4. Any concurrent respiratory disease as bronchiectasis, COPD, lung fibrosis, …
5. Current or known history of tuberculosis in any organ.
6. Current malignancy or any history of malignant disease for the past 5 years.
7. Subjects receiving any medications with known drug interaction with study medications.
8. Use of beta-blockers including eye drops.
9. Any significant concurrent disease as cardiac, hepatic, renal, …
10. Current or history of alcohol or drug abuse.
11. Current or history of significant psychiatric disease.
12. Current or history of significant immunodefieciency.
13. History of receiving any biological therapy for asthma for the last 3 years or currently eligible for any biological therapy for asthma.
14. Subjects under any immuno-modulating therapy including biological therapy for any other indication. Subjects may be allowed to participate after 5 times half-live of the concerned drug.
15. Any known allergy or contraindication to any of the study medications.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed mild to moderate asthma, aged 12 years and above, with no significant comorbidity/ies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Annualized frequency of asthma step-up | 52 weeks
  Event in which the patient is considered eligible for step-up of asthma therapy. Any of the following is considered as asthma step-up:
  1. Use of reliever medication once daily or more for successive 7 days.
  2. Use of reliever medication for 2 times or more for successive 3 days.
  3. Any severe exacerbation as per protocol definition.
  4. Increase in weekly ACQ-5 score (with higher score means worse asthma control) by 0.5 or more points.
  5. Persistent decrease in PEF by 20% or more from baseline for 3 days or more.

SECONDARY OUTCOMES:
Annualized frequency of asthma step-down. | 52 weeks
  Event in which the patient is considered eligible for step-down of asthma therapy. All of the following is required for asthma step-down:
  1. Use of reliever medications 2 times or less weekly for at least 4 successive weeks.
  2. No severe exacerbation for 12 weeks or more.
  3. ACQ-5 score of 0.5 or less persistently for 4 successive weeks or more.
  4. PEF record with a variability of 10% or less for 4 successive weeks or more.
  5. No previously recorded deterioration as per asthma step-up definition for 12 weeks or more.
Annualized rate of asthma severe exacerbation. | 52 weeks
  Continuous and/or abrupt worsening of asthma which require any of the following:
  1. Hospitalization for asthma exacerbation.
  2. ER visit with consequent administration of any form of systemic corticosteroids.
  3. Prescription of OCS for ≥3 days.
  4. Persistent decrease of PEF by 30% or more from baseline for 2 successive days or more.
Annualized rate of asthma control weeks. | 52 weeks
  Asthma control weeks is measured by asthma control questionnaire-5 (ACQ-5) weekly, with higher score means worse asthma control.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham H Raafat, M.D., Principal Investigator — Security Forces Hospital Dammam
Locations (1):
- Security Forces Hospital Dammam, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided